CLINICAL TRIAL: NCT00489164
Title: A Randomized Feasibility Study With the Sirolimus-Eluting BX Velocity Balloon-Expandable Stent in the Treatment of Diabetic Patients With Native Coronary Artery Lesions (DECODE)
Brief Title: Feasibility Study With the Sirolimus-Eluting BX Velocity Balloon-Expandable Stent in the Treatment of Diabetic Patients With Native Coronary Artery Lesions
Acronym: DECODE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P02-6316, P01-6311
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Peripheral Vascular Diseases
Keywords: DIABETIC PATIENTS WITH NATIVE CORONARY ARTERY LESIONS
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Sirolimus-Eluting BX Velocity Balloon-Expandable Stent

SUMMARY:
The main objective of this study is to assess in-stent late lumen loss in diabetic patients with de novo native coronary lesions using the sirolimus-eluting Bx VELOCITYä stent as compared to the Bx VELOCITY balloon-expandable stent.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be 18 years of age;
2. Patients must be previously diagnosed with Type I or Type II diabetes with documented treatment with insulin or oral hypoglycemics by medical history. (Undocumented or newly diagnosed diabetics must have fasting plasma glucose of >/= 126 mg/dl or a 2h post-load value in the OGTT >/=200 mg/dl, confirmed on alternate days);
3. Female of childbearing potential must have a negative pregnancy test and must plan to be on accepted method of contraception for 6 months after time of enrollment;
4. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;
5. Treatment of lesions in native coronary arteries requiring a maximum of three stents per patient. Multi-vessel treatment is permissible. Additional stents may be used for procedural complications such as dissections. Patients with additional lesions can be included only if the other lesions are not considered clinically significant and do not require treatment;
6. Target lesion is >/=2.25 and </=3.0 in diameter (visual estimate);
7. Individual lesions are >/=10 mm to </= 32 mm in length located in a native coronary artery;
8. Target lesions are de novo lesions in native coronary vessels;
9. Acceptable candidate for coronary artery bypass surgery (CABG);
10. Target lesion stenosis is >50% and <100% (TIMI I) (visual estimate);
11. Patient is willing to comply with the specified follow-up evaluation;
12. Patient must provide written informed consent prior to the procedure using a form that is approved by the local Institutional Review Board.

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK>2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remains above normal at the time of treatment;
2. Unprotected left main coronary disease with 50% stenosis;
3. Significant (>/=50%) stenoses proximal or distal to the target lesion that might require revascularization or impede runoff;
4. Patients admitted for treatment of diabetic ketoacidosis >/= 2 times in the past six months (Brittle Diabetics);
5. Intervention of another lesion has occurred within six months prior to index procedure;
6. Have an ostial target lesion;
7. Target lesion is in a saphenous venous graft.
8. Target lesion is due to in-stent restenosis.
9. Angiographic evidence of thrombus within target lesion;
10. Calcified lesions which cannot be successfully predilated;
11. Ejection fraction </=30%;
12. Totally occluded vessel (TIMI 0 level);
13. Impaired renal function (creatinine > 2.0 mg/dL);
14. Target lesion has excessive tortuosity unsuitable for stent delivery and deployment;
15. Pretreatment with devices other than balloon angioplasty (direct stenting is not allowed);
16. Target lesion involves bifurcation including a side branch >/=2.5mm in diameter (either stenosis of both main vessel and major branch or stenosis of just major branch) that would require side branch stenting which is likely to occur if side branch is diseased and intended to be stented;
17. Previous brachytherapy of target vessel;
18. Recipient of heart transplant;
19. Patient with a life expectancy less than 12 months;
20. Known allergies to aspirin, clopidogrel bisulfate (Plavix) and ticlopidine (Ticlid), heparin, stainless steel, contrast agent or sirolimus, that cannot be medically managed;
21. Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study;
22. Currently participating in an investigational drug or another device study;
23. Treatment with Metformin (glucophage) within 48 hours of angiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2002-08; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss as measured by QCA at six months post-procedure. In-stent measurement is defined as the measurement within the stented segment. | 6 months post-procedure

SECONDARY OUTCOMES:
Composite of Major Adverse Cardiac Events (MACE) defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat target lesion revascularization at 30 days, 6 months and 1 year post-procedure | at 30 days, 6 months and 1 year post-procedure
Target lesion revascularization (TLR) and target vessel revascularization (TVR) at 30 days, 6 months and 1 year post-procedure | at 30 days, 6 months and 1 year post-procedure
Target vessel failure (TVF) defined as cardiac death, myocardial infarction, or target vessel revascularization at 30 days, 6 months and 1 year post-procedure | at 30 days, 6 months and 1 year post-procedure
Device success defined as achievement of a final residual diameter stenosis of <50% (by QCA), using the assigned device only. If QCA is not available, the visual estimate of diameter stenosis is used | Throughout study
Lesion success defined as the attainment of <50% residual stenosis (by QCA) using any percutaneous method | Throughout study
Procedure success defined as achievement of a final diameter stenosis of <50% (by QCA) using any percutaneous method, without the occurrence of death, MI, or repeat revascularization of the target lesion during the hospital stay | Throughout study
In-stent mean percent diameter stenosis (%DS), Binary restenosis and late lumen loss as measured by quantitative coronary angiography at post-procedure and at 6-months | at post-procedure and at 6-months
In-lesion mean percent diameter stenosis (%DS), mean lumen diameter (MLD), binary restenosis and late lumen loss as measured by quantitative coronary angiography at post-procedure and at 6-months | at post-procedure and at 6-months
Glycemic control as measured by HbA1C at 6 months and 1 year follow-up | at 6 months and 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Buchbinder, MD, Principal Investigator — Scripps Memorial Hospital
Locations (11):
- United States (4):
  - Foundation for Cardiovascular Medicine, La Jolla, California
  - Florida Hospital, Orlando, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St Luke's Hospital, Kansas City, Missouri
- Queen Mary Hospital, Hong Kong, China
- India (4):
  - Batra Hospital & Research Centre, New Delhi, National Capital Territory of Delhi
  - Apollo Hospital, Chennai, Tamil Nadu
  - Jaslok Hospital & Research Centre, Mumbai
  - Escorts Heart Institute & Research Centre, New Delhi
- National Heart Institute, Kuala Lumpur, Malaysia
- National Heart Center, Singapore, Singapore

REFERENCES:
- [Result] Chan C, Zambahari R, Kaul U, Lau CP, Whitworth H, Cohen S, Buchbinder M; DECODE Investigators. A randomized comparison of sirolimus-eluting versus bare metal stents in the treatment of diabetic patients with native coronary artery lesions: the DECODE study. Catheter Cardiovasc Interv. 2008 Nov 1;72(5):591-600. doi: 10.1002/ccd.21719. PMID 18949772